CLINICAL TRIAL: NCT06628076
Title: Antibacterial Effect of Zinc Oxide Nanoparticles on Acinetobacter Baumannii Isolated from Patients with Hospital Acquired Infections in Sohag University Hospitals, Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shimaa Anwar Ahmed, Assistant lecturer of Medical Microbiology and Immunology, Sohag University
Other Study IDs: Soh-Med-24-9-1MD
Record Dates: First submitted 2024-09-26; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Infections, Nosocomial; Infections, Respiratory Tract
Keywords: A. baumannii.; Biofilm; ZnO NPs; hospital aquired infections
MeSH Terms: conditions — Cross Infection; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Different samples (pus, urine, urinary catheter samples, wound swabs, sputum, bronchoalveolar lavage and central venous catheter samples) will be collected under strict aseptic precautions from patients admitted at different departments at Sohag university hospitals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Culture specific antibiotic therapy — Samples will be cultured on MacConkey agar. Morphological identifications of growth isolates by Gram staining, colony features and conventional biochemical tests. All isolates will be identified to species level using automated bacterial identification systems.
Diagnostic Test: Antibiotic — Strains confirmed as A. baumannii will be examined for their different antibiotic susceptibility by modified Kirby Bauer's disc diffusion method on Mueller Hinton Agar.
Diagnostic Test: Biofilm assessment — The biofilm formation activity of A. baumannii isolates will be tested using the microtitre plate technique
Diagnostic Test: nanoparticle zinc oxide — Detection of the effect of ZnO NPs on the biofilm producer MDR A. baumannii strains using the same method
Diagnostic Test: Molecular detection of antibiotic resistance — - Evaluation the effect of ZnO NPs on the expression of some efflux pump genes, and biofilm related genes in MDR A. baumannii isolates using Real time PCR technology.

SUMMARY:
A. baumannii is known as the most frequently isolated organism in intensive care units (ICUs), causing a variety of nosocomial infections, including pneumonia, urinary tract infections (UTIs), bacteremia as well as skin and soft tissue infections. These infections are usually associated with high mortality rates ranging between 26% among hospitalized patients and 43% among ICU patients.

DETAILED DESCRIPTION:
Acinetobacter baumannii (A. baumannii) is Gram- negative, aerobic, glucose non-fermentative, non-motile coccobacillus, ubiquitous in nature, and persistent in healthcare settings. It is regarded as a significant opportunistic human pathogen.

This bacterium become a growing problem in hospitals as a predominant multidrug-resistant (MDR) bacterium. Horizontal acquisition of resistance genes is the main factor involved in the emergence of MDR .

There are many mechanisms to confer resistance to different classes of antibiotics in A. baumannii, one of them is multidrug efflux pumps. These efflux pumps are important source of MDR, which export antibiotics from the cell, increasing their antibiotic resistance.

AdeABC is one of the most important efflux systems, belonging to the RND family in Acinetobacter, which plays an important role in the resistance to a broad group of antibiotics; its genes are chromosomal and encode three genes, i.e., AdeB, AdeA, and AdeC, forming an operon in the vicinity. In addition, the expression of AdeABC is done by a two-component system, which includes a response regulator (AdeR) and a sensor kinase (AdeS) .

The ability of Acinetobacter spp. to form biofilm that enables bacterial survival in hospital settings, especially in ICUs, is the most significant contributing factor to their virulence, and this trait is also responsible for their notable antibiotic resistance. Several biofilm-related genes influence antimicrobial susceptibility, suggesting an association between the biofilm-forming ability of Acinetobacter spp. and their antibiotic resistance patterns (MDR/XDR)

Zinc oxide nanoparticles (ZnO NPs) are one of the most important nanoparticles of metal oxides; it is a unique and inorganic materials that can be used in several biological applications (anti-bacterial, anti-inflammatory). ZnO NPs exhibit distinctive properties other than other nanoparticles such as higher solubility, better biofilm penetration and effective drug delivery . ZnO NPs have been reported to have antimicrobial properties such as disrupting the cell membrane of pathogens, accumulating in the cell and producing toxic H2O2 (hydrogen peroxide)

ELIGIBILITY:
Inclusion Criteria:

* All patients suffering from infections that can be caused by A. baumannii.

Exclusion Criteria:

* All patients suffering from infections that aren't caused by A. baumannii.

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will be carried out at Department of Medical Microbiology and Immunology, Sohag Faculty of Medicine and Sohag University Hospitals.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2024-10-10 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
A. baumannii antibiotic susceptibility profile | October 2024 to December 2025
  A. baumannii antibiotic susceptibility profile will be done using modified kirbybeur method
Isolation and identification of A. baumannii from different clinical samples | October 2024 to December 2025
  Isolation and identification of A. baumannii from different clinical samples using MacConKey medium, oxidase test. TSI, And automated identification ViteK system
A. baumannii strains which produce biofilm | October 2024 to December 2025
  Detection of A. baumannii strains which produce biofilm using tissue culture plates and Gram stain
Ability of ZnO NPs to inhibit the phenomenon of biofilm formation by MDR A. baumannii strains | October 2024 to December 2025
  Assessment of ability of ZnO NPs to inhibit the phenomenon of biofilm formation by MDR A. baumannii strains using ZnO NPs to be applied by different concentrations on tissue culture plates and measure the degree of Biofilm formation using ELISA
The effect of ZnO NPs on the expression of some efflux pump genes and biofilm related genes in MDR A. baumannii strains | October 2024 to December 2025
  Evaluation the effect of ZnO NPs on the expression of some efflux pump genes and biofilm related genes in MDR A. baumannii strains using real time PCR(Polymerase Chain reaction)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://dx.doi.org/10.4103/ecdt.ecdt_40_23